CLINICAL TRIAL: NCT02689011
Title: Incidence of Urinary Retention in Patients Undergoing Unilateral Total Knee Arthroplasty- Comparison Between Continuous Epidural Analgesia and Single Shot Femoral Nerve Block- a Randomized Controlled Study (UriKANE)
Acronym: UriKANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ausaf Ahmed Khan, Resident, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CTU / UriKANE / 2013
Record Dates: First submitted 2016-02-07; First posted 2016-02-23 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Acute Pain; Urinary Retention; Post Operative Pain
Keywords: Total Knee Arthroplasty; Femoral Nerve Block; Epidural Analgesia; Urinary Retention; Lumbar Epidural
MeSH Terms: conditions — Acute Pain; Urinary Retention; Pain, Postoperative | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group F (Experimental): Femoral nerve Block Group
  Interventions: Procedure: Femoral Nerve Block
- Group E (Active Comparator): Epidural Group
  Interventions: Procedure: Epidural

INTERVENTIONS:
Procedure: Femoral Nerve Block — For patients in Femoral nerve Block Group (Group F), ultrasound guided Femoral nerve block was performed using 0.375% bupivacaine, 20 ml for femoral nerve
  Arms: Group F
Procedure: Epidural — Patients in Epidural Group (Group E) were turned in lateral position for epidural catheter placement in lumbar region. Epidural was loaded with 0.25% bupivacaine and infusion of M2 (Bupivacaine 0.1% + Fentanyl 2mcg/ml) was started at 8 - 12 ml per hour.
  Arms: Group E

SUMMARY:
This study aims to compare the incidence of urinary retention and requirement of bladder catheterization in patients undergoing total knee arthroplasty while receiving either continuous epidural analgesia or single shot femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical status I, II & III
* Male and Female Patients age between between 30 and 70 years
* Unilateral Total Knee Arthroplasty

Exclusion Criteria:

* Patient Refusal
* Allergy to local anesthetics, paracetamol or other study drugs
* History of opioid dependence
* Contraindications to spinal/epidural anesthesia and femoral nerve block (coagulation defects, infection at puncture site etc.)
* Inability to use patient-controlled analgesia (IV PCIA) (as assessed at the time of informed consent)
* History of urinary retention, neurogenic bladder, or any urologic problem

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary retention | 24 Hours
  To compare the incidence of urinary retention in patients undergoing unilateral Total Knee Arthroplasty receiving continuous epidural analgesia vs. single shot Femoral Nerve Block.

SECONDARY OUTCOMES:
Mean post-operative nausea and vomiting scores | up to 48 hours
  To compare the mean post-operative nausea and vomiting scores between the two groups at 0, 1, 12, 24 & 48 hours postoperatively.
Mean post-operative sedation scores | up to 48 hours
  To compare the mean post-operative sedation scores between the two groups at 0, 1, 12, 24 & 48 hours postoperatively.
Mean post-operative pain scores | up to 48 hours
  To compare the mean post-operative pain scores between the two groups at 0, 1, 12, 24 & 48 hours postoperatively.
Surgical outcomes - maximal knee flexion | up to 48 hours
  To compare surgical outcomes like maximal knee flexion at 24 & 48 hours between the two groups
Surgical outcomes - duration of post-operative hospital stay | up to 48 hours
  To compare surgical outcomes like duration of post-operative hospital stay between the two groups
Surgical outcomes - mobilization out of bed | up to 48 hours
  To compare surgical outcomes like time taken to mobilize out of bed between the two groups
Surgical outcomes - food intake | up to 48 hours
  To compare surgical outcomes like time of first food intake between the two groups
Patient satisfaction | 7 Days
  To compare Patient satisfaction with the analgesic modality between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ausaf A Khan, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes